CLINICAL TRIAL: NCT06207071
Title: Early DHA Supplementation in Growth-restricted Very Preterm Infants: A Randomized Clinical Trial
Brief Title: Early DHA/ARA Supplementation in Growth-restricted Very Preterm Infants: A Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Mead Johnson Nutrition (Industry)
Responsible Party: Principal Investigator, Ariel A. Salas, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 300012038
Record Dates: First submitted 2024-01-05; First posted 2024-01-16 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Infant Malnutrition; Light-For-Dates With Signs of Fetal Malnutrition; Premature; Nutrition Disorder, Infant
MeSH Terms: conditions — Infant Nutrition Disorders; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): A DHA/ARA supplement will be added to expressed human milk or donor human milk administered during the first 3 weeks after birth.
  Interventions: Dietary Supplement: DHA
- Control (No Intervention): No DHA/ARA supplement will be added to expressed human milk or donor human milk administered during the first 3 weeks after birth.

INTERVENTIONS:
Dietary Supplement: DHA — DHA supplementation
  Arms: Intervention

SUMMARY:
Growth-restricted very preterm infants (VPT) are born without adequate fat mass (FM) deposits and low docosahexaenoic acid (DHA) concentrations. They often experience further declines in DHA concentrations during the initial three weeks post-birth while advancing enteral feeds and receiving lipid supplementation predominantly through parenteral nutrition. These suboptimal enteral and parenteral nutrition practices significantly heighten the risk of faltering postnatal growth. One promising approach to mitigate these issues is enteral DHA supplementation. However, it remains unclear whether the early administration of DHA through enteral supplementation could lead to a more substantial increase in head growth without affecting FM accretion in growth-restricted VPT infants. To address this question, we propose a masked randomized clinical trial involving 152 VPT infants.

ELIGIBILITY:
Inclusion Criteria:

* Gestational ages between 22 0/7 - 32 6/7 weeks gestation
* < 25th centile birthweight

Exclusion Criteria:

* Major congenital/chromosomal anomalies
* Terminal illness in which decisions to withhold or limit support have been made

Ages: 24 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Head circumference at 36 weeks postmenstrual age or discharge | Birth to 36 weeks postmenstrual age or discharge
  Declines in head circumference z scores from birth to 36 weeks postmenstrual age

SECONDARY OUTCOMES:
Fat mass(FM)-for-age Z-score | Birth to 36 weeks postmenstrual age
  FM accretion will be estimated by air displacement plethysmography
Changes in serum metabolic profile at 36 weeks postmenstrual age | 36 weeks postmenstrual age or discharge
  Determined by metabolomic analyses of serum samples

OTHER OUTCOMES:
Cognitive outcomes | 2 years of age
  Determined by Bayley assessment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States